CLINICAL TRIAL: NCT04947163
Title: Effects of Inspiratory Muscle Training (IMT) on Balance Ability and Quality of Life of Diabetes Mellitus Patients
Acronym: IMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/13564 Suman Sheraz
Record Dates: First submitted 2021-06-26; First posted 2021-07-01 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus
Keywords: Balance; Diabetes Mellitus; Inspiratory Muscle Training; Quality of life
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IMT group (Experimental): * Standard exercise protocol according to ACSM's guidelines Standard exercise protocol according to ACSM's guidelines
  * Balance training - Otago Exercise Program (OEP)
    * warm-up (10-15 min)
    * strengthening exercises (~20 min)
    * balance activities (~20 min)
    * cool-down (5-10 min) Balance training - OEP
    * warm-up (10-15 min)
    * strengthening exercises (~20 min)
    * balance activities (~20 min)
    * cool-down (5-10 min)
  * IMT through POWERBREATHE
    * 30 quick breaths twice daily at an adjustable resistance (equivalent to ~50% of [baseline] MIP).
    * Will be increased up to 35 breaths as per patient's tolerance Sham IMT
    * 60 slow breaths once daily at a load setting of 0 (corresponding to ~15% [baseline] MIP)
    * training load adjustment will be prevented using sticky tape applied to the device's load adjuster.
  Interventions: Device: Inspiratory Muscle Training
- Sham IMT (Sham Comparator): * Standard exercise protocol according to ACSM's guidelines Standard exercise protocol according to ACSM's guidelines
  * Balance training - OEP
    * warm-up (10-15 min)
    * strengthening exercises (~20 min)
    * balance activities (~20 min)
    * cool-down (5-10 min) Balance training - OEP
    * warm-up (10-15 min)
    * strengthening exercises (~20 min)
    * balance activities (~20 min)
    * cool-down (5-10 min)
  * IMT through POWERBREATHE
    * 30 quick breaths twice daily at an adjustable resistance (equivalent to ~50% of [baseline] MIP).
    * Will be increased up to 35 breaths as per patient's tolerance Sham IMT
    * 60 slow breaths once daily at a load setting of 0 (corresponding to ~15% [baseline] MIP)
    * training load adjustment will be prevented using sticky tape applied to the device's load adjuster.
  Interventions: Device: Sham IMT

INTERVENTIONS:
Device: Inspiratory Muscle Training — Participants will perform home-based IMT twice daily [once in the morning (between 7:00 and 12:00 am) and once in the evening (between 16:00 and 21:00 pm)], for 8 consecutive weeks, using a mechanical pressure threshold loading device. In addition, participants in this group will try to increase the inspiratory resistance when the participants feel that 30 breaths are achievable with ease or if the participants could reach 35 consecutive breaths.
  Arms: IMT group
Device: Sham IMT — Participants will perform 60 slow breaths once daily at a load setting of 0 (corresponding to ~15% [baseline] MIP), using the same device as the IMT group. For the sham group, the ability to adjust the training load will be prevented using sticky tape applied to the device's load adjuster.
  Arms: Sham IMT

SUMMARY:
The disease burden of Diabetes Mellitus (DM) is growing rapidly, and multiple complications have been reported including cardiopulmonary and high fall risk which declines the overall quality of life. IMT can be useful technique to improve the physical and functional performance, reduce the severity of complications and enable the individuals to become active members of community. The current study is intended to evaluate the dual effects of IMT on postural stability and pulmonary function of diabetic patients.

DETAILED DESCRIPTION:
Diabetes Mellitus (DM) is a chronic metabolic disease characterized by hyperglycemia due to either deficiency of insulin or the inability of the body to utilize it. Hyperglycemia ultimately leads to multiple organ damage in patients with uncontrolled diabetes. The incidence occurs mostly at the age of 55 years equally affecting both genders. The prevalence of diabetes has been increased four times in the last three decades worldwide and global prevalence is increasing alarmingly with about 1 out of every 11 individuals having diabetes mellitus with 90% patients having type 2 diabetes mellitus. The statistical data depicts a huge burden of disease both in morbidity and mortality globally and an anticipated threat on health care system in future. (1) The complications of diabetes have been reported higher in the South Asia region as compared to western counterparts. In Pakistan, according to National Diabetes Survey of Pakistan (NDSP 2016 - 2017), the pooled prevalence of diabetes was projected to be 26.3% affecting 27.4 million people above 20 years of age. These high numbers are directly and indirectly linked with the economic burden on society and ultimately affect the quality of life of diabetics, families, and community.

Clinically, there are different complications (micro & macro vascular) associated with DM and these are main sources of morbidity and mortality. Neuropathy, nephropathy, and retinopathy are the microvascular complications whereas macrovascular complications include cardiovascular diseases, stroke as well as other vascular diseases. Apart from these complications, there are few other complications including decreased resistance to infections, dental issues, birth complications in gestational diabetes, poor balance, sarcopenia and increased risk of fall and fractures. The reduced strength and endurance of diaphragm the vital muscle of respiration lead to compromised respiratory functions.

Peripheral neuropathy, retinopathy and vestibular impairments alter the biomechanical stability and strength of postural control in individuals with DM. The instability generates disparity among muscular and neural structures to execute locomotion abilities, so abnormal gait pattern, weakness in lower limb musculature, impair sensory function, diminished reflexes and high fall risk have been observed.

These musculoskeletal complications compromise the mobility level and impede the performance of functional tasks and Activities of Daily Life (ADLs) in patients with DM. The limited movements and participation restrictions in social activities create inaccessibility and dependence on caregiver has been increased. The overall activity level has been declined and decreases the quality of life of individuals and ultimately developing social and economic burden on community.

Management of DM always emphases to improve the current health status and prevent further complications due to uncontrolled DM. Multiple management approaches have been reported in the literature to maintain adequate glycemic control and manage diabetes related complications and co morbidities. Treatment strategies also focus to maximize the quality of life and minimize the risk of treatment related complications including hypoglycemia. Balance and postural impairments are common in DM due to neuropathic changes and there are different training strategies have been documented in literature to improve postural stability and reduce fall risk. The training approaches include Tai Chi, Wii Fit based training, circuit training, strengthening exercises of lower limbs, gait training and task oriented dynamic training to enhance the overall balance abilities.

The central trunk stability and core strength are integral part of postural stability and balance but there is limited evidence to address these for balance training in DM. There is lacking evidence in literature on specific training targeting the central trunk and core strength to improve the balance ability, reduces fall risk and improve quality of life in DM patients.

Inspiratory Muscle Training (IMT) is a device-based training and widely used therapeutic technique for improving inspiratory muscle strength and endurance, thoracic mobility, exercise capacity, reducing dyspnea and increasing quality of life. Recently, IMT has been used to improve balance and physical performance among elderly.

How IMT is a useful intervention to improve cardiopulmonary function, postural control and quality of life? The underlying mechanism of IMT principal and clinical implications has three-fold mechanisms:

First: Diaphragm thickness and strength enhances balance in two ways. Firstly, there is activation of diaphragm during upper limb movements indicating that the co-activation of diaphragm assists in the mechanical stabilization of the spine. Secondly, it plays a major role in the generation of intra-abdominal pressure which helps in the stabilization of lumbar spine during movements like shoulder abduction and adduction i.e., balance perturbations. These changes will improve the lower limb mobility, quadriceps strength, functional performance, postural control response and exercise tolerance among individuals. It creates an overall impact on enhanced balance strategies, physical performance and postural stability in elderly and other pathological conditions including chronic obstructive pulmonary disease (COPD), cystic fibrosis and stroke.

Second: Increases in diaphragmatic mobility and hypertrophy as well as improved neural control and thickness of respiratory muscles including transversus abdominus and internal obliques leads to increase in exercise capacity, pulmonary function and decreased perceived breathlessness and exertion in the patients. It will increase the strength of respiratory muscles ultimately proving it to be an effective treatment strategy in COPD, chronic heart failure, multiple sclerosis and various respiratory diseases.

Third: IMT exerts certain ergogenic effects through increasing diaphragmatic mobility and strength thereby improving the recovery time in sprinters, limiting cardiac sympathetic hyperactivity in cyclists and enhance rowing performance.

Therefore, it can be hypothesized that IMT is not only effective for improving cardiopulmonary function but is also strongly linked with postural stability. The disease burden of DM is growing rapidly, and multiple complications have been reported including cardiopulmonary and high fall risk which declines the overall quality of life. IMT can be useful technique to improve the physical and functional performance, reduce the severity of complications and enable the individuals to become active members of community. The current study is intended to evaluate the dual effects of IMT on postural stability and pulmonary function of diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Mini Mental State Examination (MMSE) score >24
* Type II diabetes: Post 5-8 years diagnosis
* Berg Balance score (30-40)
* Presence of polyneuropathy confirmed through Modified Toronto Clinical Scoring System.

Exclusion Criteria:

* Patients on oxygen therapy
* Uncontrolled diabetes (Confirmed through HbA1C) or disease exacerbation in last 3 months.
* Patients practicing regular physical activity, any balance training in the last 6 months and previous or current experience with IMT
* Patients with musculoskeletal comorbidities that may impair exercise performance
* Peripheral oxygen saturation (SpO2) < 90% during the Six-Minute Walk Test (6MWT)
* Patients with long COVID syndrome
* Hypertensive subjects without control medication as well as those presenting with a hypertensive peak (> 140/90 mmHg) for more than 3 consecutive days
* Patients with cardiorespiratory diseases or patients taking drugs that effect balance e.g., beta blockers, anti-anxiety and anti-depressant drugs.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Fall risk score | After 12 weeks of intervention
  Fall risk score will be calculated by Biodex Postural Stability system which is a highly reliable and objective measure for assessment of balance. It provides a 20o surface tilt in all 360 degree directions while providing an adjustable spring resistance to mobile surface from a static base of support at level 12 to a fully mobile base of support of level 1 same as wobble board like movements. Higher scores of fall risk score indicate greater balance deterioration and thus increase risk of fall. It would be assessed at baseline, after 12 weeks and after 6months of intervention.
Overall stability index | After 12 weeks of intervention
  Overall stability index will be calculated through Biodex Postural Stability system which is a highly reliable and objective measure for assessment of balance. It provides a 20o surface tilt in all 360 degree directions while providing an adjustable spring resistance to mobile surface from a static base of support at level 12 to a fully mobile base of support of level 1 same as wobble board like movements. It would be assessed at baseline, after 12 weeks and after 6months of intervention.
Anterior / Posterior index | After 12 weeks of intervention
  Anterior / Posterior index will be calculated through Biodex Postural Stability system which is a highly reliable and objective measure for assessment of balance. It provides a 20o surface tilt in all 360 degree directions while providing an adjustable spring resistance to mobile surface from a static base of support at level 12 to a fully mobile base of support of level 1 same as wobble board like movements. It would be assessed at baseline, after 12 weeks and after 6months of intervention.
Medial / lateral index | After 12 weeks of intervention
  Medial / lateral index will be calculated through Biodex Postural Stability system which is a highly reliable and objective measure for assessment of balance. It provides a 20o surface tilt in all 360 degree directions while providing an adjustable spring resistance to mobile surface from a static base of support at level 12 to a fully mobile base of support of level 1 same as wobble board like movements. It would be assessed at baseline, after 12 weeks and after 6months of intervention.
Modified Clinical Test of Sensory Interaction in Balance (M - CTSIB) (composite score) | After 12 weeks of intervention
  Modified Clinical Test of Sensory Interaction in Balance (M - CTSIB) will be calculated through Biodex Postural Stability system which is a highly reliable and objective measure for assessment of balance. It provides a 20o surface tilt in all 360 degree directions while providing an adjustable spring resistance to mobile surface from a static base of support at level 12 to a fully mobile base of support of level 1 same as wobble board like movements. It would be assessed at baseline, after 12 weeks and after 6months of intervention.
Audit of Diabetes Dependent Quality of Life: | After 12 weeks of intervention
  Audit of Diabetes Dependent Quality of Life (ADDQOL) is a reliable questionnaire used to measure individual's perception of the impact of diabetes on their quality of life. The scales range from -3 to +1 for 19 life domains (impact rating) and from 0 to +3 in attributed importance (importance rating). A weighted score for each domain is calculated as a multiplier of impact rating and importance rating (ranging from -9 to +3). Lower scores reflect poorer quality of life. It would be assessed ay baseline, after 12 weeks and after 6months of intervention.

SECONDARY OUTCOMES:
Peak expiratory flow rate (PEFR) | After 12 weeks of intervention
  Peak expiratory flow rate (PEFR) measured through digital spirometer. Peak Expiratory Flow Rate (PEFR) measured through digital spirometer. Three zones of measurement are commonly used to interpret peak flow rates. Normal value of PEFR is (80-100%). Green zone indicates 80 to 100 percent of the usual or normal peak flow reading, yellow zone indicates 50 to 79 percent of the usual or normal peak flow readings, and red zone indicates less than 50 percent of the usual or normal peak flow readings. It would be assessed at baseline, after 4th, 8th and 12th weeks of intervention.
Forced vital capacity (FVC) | After 12 weeks of intervention
  Forced vital capacity (FVC) measured through digital spirometer. If the value of FVC is within 80% of the reference value, the results are considered normal. It would be assessed at baseline, after 4th, 8th and 12th weeks of intervention.
Forced expiratory volume in 1sec (FEV1) | After 12 weeks of intervention
  Forced expiratory volume in 1sec (FEV1) measured through digital spirometer. If the value of FEV1 is within 80% of the reference value, the results are considered normal. It would be assessed at baseline, after 4th, 8th and 12th weeks of intervention.
FVC/FEV1 | After 12 weeks of intervention
  FVC/FEV1 measured through digital spirometer. The normal value for the FEV1/FVC ratio is 70% (and 65% in persons older than age 65). It would be assessed at baseline, after 4th, 8th and 12th weeks of intervention.
Biering-Sørensen tests | After 12 weeks of intervention
  Posterior trunk muscle endurance will be assessed using the Biering-Sørensen test, where participants will be asked to maintain a prone position, facing the floor, with their torso unsupported over the edge of the test bench. A strap will secure their legs and hips, and hands will be placed behind their head. It would be assessed at baseline, after 4th, 8th and 12th weeks of intervention.
Sit up test | After 12 weeks of intervention
  Anterior trunk muscle endurance will be assessed using an isometric 'sit-up' task, by adopting a bent knee (~75°) sit-up. A strap will secure participants' feet, their arms will be folded across the chest, while their back will be placed against a support (60° angle from the testbed), and knees and hips will be flexed to 90 degree. It would be assessed at baseline, after 4th, 8th and 12th weeks of intervention.
Six Minute Walk test (6MWT) | After 12 weeks of intervention
  Six Minute Walk test (6MWT) will be used to assess the functional capacity of the patients. The subjects will be instructed to walk for 6 minutes at a given time along a 30-m line at an interval of 1.5 m in an outdoor corridor, and the distance walked will be recorded in meters. The patients will be encouraged to continue walking as fast as possible. It would be assessed at baseline, after 4th, 8th and 12th weeks of intervention.
30sec sit-to-stand (30secSTS) | After 12 weeks of intervention
  30sec sit-to-stand (30secSTS) is a test of physical performance which involves measuring the number of times participants can stand from a seated position, and then become seated again in 30 second period. ( Participants will be asked to sit on the edge of an armless chair (sitting height 46 cm, seat length 45 cm) with their arms folded across their chest. Participants will be instructed to rise, and then become seated as fast as possible, and as many times as possible in 30 seconds, with both feet maintaining contact with the floor at all time. It would be assessed at baseline, after 4th, 8th and 12th weeks of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Nawaz Malik, PhD, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway Hospital, Riphah Rehabilitation Center, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized, individual participant data that underlie results reported in this article will be shared on request (at suman.sheraz@riphah.edu.pk) as an excel file immediately after publication till 36 months of publication as per policy of university. Later on it will be available on university repository. Study protocol and analysis plan are also shared as supplementary files.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication till 36months
Access Criteria: on reasonable request

REFERENCES:
- [Background] Mustapa A, Justine M, Mohd Mustafah N, Jamil N, Manaf H. Postural Control and Gait Performance in the Diabetic Peripheral Neuropathy: A Systematic Review. Biomed Res Int. 2016;2016:9305025. doi: 10.1155/2016/9305025. Epub 2016 Jul 20. PMID 27525281
- [Background] Ferraro FV, Gavin JP, Wainwright T, McConnell A. The effects of 8 weeks of inspiratory muscle training on the balance of healthy older adults: a randomized, double-blind, placebo-controlled study. Physiol Rep. 2019 May;7(9):e14076. doi: 10.14814/phy2.14076. PMID 31074198
- [Background] Chapman A, Meyer C, Renehan E, Hill KD, Browning CJ. Exercise interventions for the improvement of falls-related outcomes among older adults with diabetes mellitus: A systematic review and meta-analyses. J Diabetes Complications. 2017 Mar;31(3):631-645. doi: 10.1016/j.jdiacomp.2016.09.015. Epub 2016 Sep 30. PMID 27765575
- [Background] Pfalzer L, Fry D. Effects of a 10-week inspiratory muscle training program on lower-extremity mobility in people with multiple sclerosis: a randomized controlled trial. Int J MS Care. 2011 Spring;13(1):32-42. doi: 10.7224/1537-2073-13.1.32. PMID 24453703
- [Background] Rodrigues GD, Gurgel JL, Galdino IDS, da Nobrega ACL, Soares PPDS. Inspiratory muscle training improves cerebrovascular and postural control responses during orthostatic stress in older women. Eur J Appl Physiol. 2020 Oct;120(10):2171-2181. doi: 10.1007/s00421-020-04441-2. Epub 2020 Jul 23. PMID 32705393
- [Background] Shei RJ, Chapman RF, Gruber AH, Mickleborough TD. Inspiratory muscle training improves exercise capacity with thoracic load carriage. Physiol Rep. 2018 Feb;6(3):e13558. doi: 10.14814/phy2.13558. PMID 29424007
- [Background] Oh D, Kim G, Lee W, Shin MM. Effects of inspiratory muscle training on balance ability and abdominal muscle thickness in chronic stroke patients. J Phys Ther Sci. 2016 Jan;28(1):107-11. doi: 10.1589/jpts.28.107. Epub 2016 Jan 30. PMID 26957739
- [Background] Gomes Neto M, Ferrari F, Helal L, Lopes AA, Carvalho VO, Stein R. The impact of high-intensity inspiratory muscle training on exercise capacity and inspiratory muscle strength in heart failure with reduced ejection fraction: a systematic review and meta-analysis. Clin Rehabil. 2018 Nov;32(11):1482-1492. doi: 10.1177/0269215518784345. Epub 2018 Jul 9. PMID 29984598
- [Background] Fry DK, Pfalzer LA, Chokshi AR, Wagner MT, Jackson ES. Randomized control trial of effects of a 10-week inspiratory muscle training program on measures of pulmonary function in persons with multiple sclerosis. J Neurol Phys Ther. 2007 Dec;31(4):162-72. doi: 10.1097/NPT.0b013e31815ce136. PMID 18172412
- [Background] Ferraro FV, Gavin JP, Wainwright TW, McConnell AK. Comparison of balance changes after inspiratory muscle or Otago exercise training. PLoS One. 2020 Jan 24;15(1):e0227379. doi: 10.1371/journal.pone.0227379. eCollection 2020. PMID 31978126
- [Derived] Sheraz S, Malik AN, Ferraro FV, Siddiqi FA. Does multifactorial inspiratory muscle training improve postural stability and quality of life of patients with diabetes in Pakistan? A randomised controlled trial. BMJ Open. 2024 Sep 16;14(9):e080718. doi: 10.1136/bmjopen-2023-080718. PMID 39284701